CLINICAL TRIAL: NCT04758481
Title: Consolidation Conventional Radiotherapy + Stereotactic Body Radiotherapy of All Body Locations With the Disease at 3 Months After First Line Chemotherapy in Stage IV Oligometastatic Non-small Cell Lung Cancer, Prior to Maintenance Therapy
Brief Title: Consolidation Conventional Radiotherapy + Stereotactic Body Radiotherapy at 3 Months After First-line Chemotherapy in Stage IV Oligometastatic Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVO-FNOs/2020-22
Record Dates: First submitted 2021-02-04; First posted 2021-02-17 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; stereotactic body radiotherapy; CyberKnife; maintenance radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is a non-randomised study with the primary intent to treat patients with NSCLC
Masking Description: The study is open label, no masking is being used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary tumour radiotherapy + stereotactic body radiotherapy + maintenance radiotherapy (Experimental): The patients, in whom disease stabilisation/partial regression will be achieved, will undergo primary tumour radiotherapy and stereotactic body radiotherapy, followed with maintenance radiotherapy.
  Interventions: Radiation: primary tumour radiotherapy; Radiation: stereotactic body radiotherapy; Radiation: maintenance radiotherapy

INTERVENTIONS:
Radiation: primary tumour radiotherapy — The study subjects will undergo primary tumour radiotherapy.
Radiation: stereotactic body radiotherapy — The study subjects will undergo stereotactic body radiotherapy.
Radiation: maintenance radiotherapy — The study subjects will undergo maintenance radiotherapy.

SUMMARY:
Lung cancer is the main cause of death among cancer diseases, in the Czech Republic, as well as worldwide. Non-small cell lung cancer (NSCLC) is responsible for more than 80% of deaths among cancer patients. Bronchogenic carcinoma is the reason of death of almost 5.500 cases every year in the Czech Republic, the mortality/incidence ration varies around 85%. The main cause for these unfavorable findings is the late detection of the carcinoma in late stages only (III and IV), when a long-term control of the disease is exceptional. Chemotherapy is able to prolong the life of patients with NSCLC by less than one year on average, that is why new treatment approaches are being examined.

DETAILED DESCRIPTION:
The basic treatment modality of lung cancer is radiotherapy, which has a proven therapeutic benefit in radical and palliative indications in up to 76% of all patients. Stereotactic robotic radiotherapy reaches maximum precision due to the precise definition of the target volume. In some localities, management with images has been solved using modern software instruments, which are able to visualize the tumor and monitor it during the whole course of respiratory cycle. This is directly associated with minimizing radiation of healthy tissues, especially the healthy lung parenchyma. In order to define predictive factors of survival of cancer patients, it is necessary to use molecular markers.

The aim of the study is to verify the feasibility of consolidation SBRT (Stereotactic Body RadioTherapy) - CyberKnife, with subsequent maintenance chemotherapy in patients with stage IV NSCLC, with max. 10 metastatic nidi. The main focus of the study will be on assessment of combination treatment toxicity.

The project is a phase I/II non-randomized clinical trial. Patients with stage IV NSCLC will be treated with 2-4 cycles of chemotherapy - platinum doublet (cisplatinum - cDDP/carboplatinum - CBDCA + Pemetrexed/navelibne - NVB). In cases when disease stabilization (SD)/partial resection (PR) will be achieved, based upon restaging examinations (CT), radiotherapy (RT) of the primary tumour will follow, with lymphadenopathy and SBRT of all metastatic nidi (max. 10 intra- or extracranial metastases). Standard fractionation schemes for RT and SBRT will be used (RT 40-50 Gy/16-20 fractions, SBRT 30 Gy/1 fractionation, 50-60 Gy/3-5 fractionations). At 3-6 weeks after the end of RT, maintenance treatment will be initiated in all patients treated with Peterexed. Regular restaging examinations are planned every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated, non-resectable, stage IV NSCLC verified with histology or cytology (according to American Joint Committee on Cancer Version 8).
* Patients must undergo 2-4 cycles of first-line chemotherapy, with the effect of disease stabilization or partial response.
* Patients over 18 years of age.
* Patients with measureable disease (on CT, PET/CT, MRI).
* Patients with 3-10 extracranial/intracranial lesions confirmed on CT, PET/CT, MRI, max. 4 weeks prior to start of SBRT.
* Max. 10 irradiated volumes (primary tumour + lymphadenopathy in one volume, if technically feasible).
* Performance status (PS) 0-2 according to ECOG. Assessment of PS max. 7 days prior to start of treatment.
* AST, ALT & ALP ≤ 2.5x norm. Total bilirubin must be within the normal range. 9. Normal function of bone marrow - Adiponectin ≥ 1.5, Haemoglobin ≥ 100, thrombo ≥ 100.
* Serum creatinine ≤1.5x norm.
* The entry laboratory tests must not be older than 14 days prior to start of treatment.
* Negative pregnancy test and use of contraception in women of childbearing age.
* Patients undergoing SBRT for pulmonary nidi must undergo entry spirometry with the value FEV1 (forced expiratory volume in 1 second) ≥ 1L.
* Patients must sign informed consent.

Exclusion Criteria:

* Patients with small-cell lung cancer or with mixed aetiology with SCLC.
* Serious ongoing infections.
* Patients with a history of haematopoiesis disorders.
* Weight loss exceeding 10% within the last 3 months.
* Patients with skin metastases of NSCLC.
* Patients treated for other malignity within the last 5 years
* Patients with more than 10 extracranial/intracranial metastases.
* Malignant fluidothorax > 1 cm prior to start of treatment.
* Patients treated with targeted treatment for EGFR mutation or EML-4-ALK translocation in the 1st-line (Erlotinib, Gefitinib, Afatinib, Crizotinib, …).
* Patients treated with immunotherapy (anti-PD-1, anti-PD-L1 or anti-PD-L2, anti CTLA-4, …).
* Participation in another clinical trial within the last month before the start of NSCLC treatment.
* Inability to cooperate or comply with the study protocol.
* Decision of the patient to discontinue participation in the study.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute and late toxicity | every 3 months, throughout the study duration, up to 32 months in total
  Acute and late toxicity of the combination therapy will be observed (according to Common Terminology for Clinical Adverse Event (CTCAE, version 5)
Progression-free survival | every 3 months
  Progression-free survival will be observed

SECONDARY OUTCOMES:
Overall survival | every 3 months, throughout the study duration, up to 32 months in total
  Overall survival will be observed
Share of nidi under local control | every 3 months, throughout the study duration, up to 32 months in total
  The share of nidi under local control will be observed (in per cent/total number of nidi)
Time to new nidus formation | every 3 months, throughout the study duration, up to 32 months in total
  The time to new nidus formation will be observed
Duration of maintenance chemotherapy | every 3 months, throughout the study duration, up to 32 months in total
  The duration of maintenance chemotherapy will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Tereza Paračková, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data with other researchers; the data may be provided upon request.

REFERENCES:
- [Background] Siva S, MacManus M, Ball D. Stereotactic radiotherapy for pulmonary oligometastases: a systematic review. J Thorac Oncol. 2010 Jul;5(7):1091-9. doi: 10.1097/JTO.0b013e3181de7143. PMID 20479693
- [Background] Onishi H, Shirato H, Nagata Y, Hiraoka M, Fujino M, Gomi K, Karasawa K, Hayakawa K, Niibe Y, Takai Y, Kimura T, Takeda A, Ouchi A, Hareyama M, Kokubo M, Kozuka T, Arimoto T, Hara R, Itami J, Araki T. Stereotactic body radiotherapy (SBRT) for operable stage I non-small-cell lung cancer: can SBRT be comparable to surgery? Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1352-8. doi: 10.1016/j.ijrobp.2009.07.1751. Epub 2010 Jul 16. PMID 20638194
- [Background] Takeda A, Kunieda E, Ohashi T, Aoki Y, Koike N, Takeda T. Stereotactic body radiotherapy (SBRT) for oligometastatic lung tumors from colorectal cancer and other primary cancers in comparison with primary lung cancer. Radiother Oncol. 2011 Nov;101(2):255-9. doi: 10.1016/j.radonc.2011.05.033. PMID 21641064
- [Background] Collen C, Christian N, Schallier D, Meysman M, Duchateau M, Storme G, De Ridder M. Phase II study of stereotactic body radiotherapy to primary tumor and metastatic locations in oligometastatic nonsmall-cell lung cancer patients. Ann Oncol. 2014 Oct;25(10):1954-1959. doi: 10.1093/annonc/mdu370. Epub 2014 Aug 11. PMID 25114022
- [Background] Norihisa Y, Nagata Y, Takayama K, Matsuo Y, Sakamoto T, Sakamoto M, Mizowaki T, Yano S, Hiraoka M. Stereotactic body radiotherapy for oligometastatic lung tumors. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):398-403. doi: 10.1016/j.ijrobp.2008.01.002. Epub 2008 Apr 18. PMID 18374506
- [Background] Guerrero E, Ahmed M. The role of stereotactic ablative radiotherapy (SBRT) in the management of oligometastatic non small cell lung cancer. Lung Cancer. 2016 Feb;92:22-8. doi: 10.1016/j.lungcan.2015.11.015. Epub 2015 Dec 2. PMID 26775592
- [Background] Oh D, Ahn YC, Seo JM, Shin EH, Park HC, Lim DH, Pyo H. Potentially curative stereotactic body radiation therapy (SBRT) for single or oligometastasis to the lung. Acta Oncol. 2012 May;51(5):596-602. doi: 10.3109/0284186X.2012.681698. Epub 2012 May 1. PMID 22548366
- [Background] Singh D, Chen Y, Hare MZ, Usuki KY, Zhang H, Lundquist T, Joyce N, Schell MC, Milano MT. Local control rates with five-fraction stereotactic body radiotherapy for oligometastatic cancer to the lung. J Thorac Dis. 2014 Apr;6(4):369-74. doi: 10.3978/j.issn.2072-1439.2013.12.03. PMID 24688781
- [Background] Lussier YA, Xing HR, Salama JK, Khodarev NN, Huang Y, Zhang Q, Khan SA, Yang X, Hasselle MD, Darga TE, Malik R, Fan H, Perakis S, Filippo M, Corbin K, Lee Y, Posner MC, Chmura SJ, Hellman S, Weichselbaum RR. MicroRNA expression characterizes oligometastasis(es). PLoS One. 2011;6(12):e28650. doi: 10.1371/journal.pone.0028650. Epub 2011 Dec 13. PMID 22174856
- [Background] Wong AC, Watson SP, Pitroda SP, Son CH, Das LC, Stack ME, Uppal A, Oshima G, Khodarev NN, Salama JK, Weichselbaum RR, Chmura SJ. Clinical and molecular markers of long-term survival after oligometastasis-directed stereotactic body radiotherapy (SBRT). Cancer. 2016 Jul 15;122(14):2242-50. doi: 10.1002/cncr.30058. Epub 2016 May 20. PMID 27206146